CLINICAL TRIAL: NCT04515667
Title: Mindfulness in the OR: Can an Abbreviated Mindfulness Skill Improve a Surgeon's Focus, Anxiety and Performance in the OR?
Brief Title: Mindfulness in the OR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HM20018279
Record Dates: First submitted 2020-08-13; First posted 2020-08-17 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Performance at Work
MeSH Terms: interventions — Mindfulness; Videotape Recording

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness (Experimental)
  Interventions: Behavioral: Mindfulness
- Control (Placebo Comparator)
  Interventions: Behavioral: Video

INTERVENTIONS:
Behavioral: Mindfulness — Participants will view a brief mindfulness video
  Arms: Mindfulness
Behavioral: Video — Participants will view a control video
  Arms: Control

SUMMARY:
The purpose of this research study is to understand the effect of a short mindfulness video on self perceived performance in the OR. Specifically, assessing the effectiveness of brief mindfulness intervention on physician focus, anxiety and perceived performance at the time of a procedure through a survey containing a modified flow state scale and modified applied mindfulness process scale

ELIGIBILITY:
Inclusion Criteria:

* practicing physicians or medical trainees
* employed in a hospital setting
* providing surgeries in an operating room setting.

Exclusion Criteria:

• practitioners involved in counseling roles

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-02-07 (Actual)

PRIMARY OUTCOMES:
Perceived flow | At the end of the procedure, up to 5 hours
  Perceived flow will be assessed using a modified flow state scale after case. Items are rated from Strongly disagree to Strongly agree. Items are summed and scored.

SECONDARY OUTCOMES:
Perceived application of mindfulness | at the end of the procedure, up to 5 hours
  Perceived mindfulness will be assess using a modified applied mindfulness process scale. Items are rated never, rarely, sometimes, often and always. Items are summed and scored.

CONTACTS AND LOCATIONS:
Overall Officials: Frances Casey, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No